CLINICAL TRIAL: NCT05383040
Title: Comparison of Percutaneous Release and Local Steroid Injection for the Treatment of Trigger Fingers: A Randomized Clinical Trial
Brief Title: Percutaneous Release vs Steroid Injection for Trigger Finger
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Armed Police Force Hospital, Nepal (Other Government)
Responsible Party: Principal Investigator, Dev Ram Sunuwar, Dietitian/Researcher, Armed Police Force Hospital, Nepal
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Trigger finger
Record Dates: First submitted 2022-05-17; First posted 2022-05-19 (Actual); Last update posted 2023-02-27 (Actual); Status verified 2023-02

CONDITIONS: Trigger Finger
Keywords: Trigger fingers; Trigger digits; Steroid injection; Percutaneous release
MeSH Terms: conditions — Trigger Finger Disorder

STUDY DESIGN:
Intervention Model Description: A hospital-based randomized clinical trial study will be carried out to compare the effect of percutaneous release of A1 pulley with steroid injection in the treatment for trigger finger.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- percutaneous release (Experimental): Percutaneous release of A1 pulley release will be performed in the well-managed operation theater set up, using an 18 gauge hypodermic needle, after preparation of the skin and injection of 1ml 2% plain lidocaine. The proper location of the pulley will be defined using surface landmarks in each digit after waiting a few minutes to allow the anesthetic to take effect the 18 gauge needle will be longitudinally moved to keep the level of the needle parallel with the tendon grating sensation will be elucidated confirming the cut of pulley until there is no grating sensation felt and improvement of symptoms. A sterile dressing will be placed.
  Interventions: Procedure: Percutaneous release
- Steroid injection (No Intervention): The steroid injection mixed with 1 ml of methyl prednisone (40mg) with 0.5 ml of 2% plain lidocaine will be inserted into the flexor tendon sheath over the A1 pulley, which will also be performed in the operation theater for patient safety.

INTERVENTIONS:
Procedure: Percutaneous release — Percutaneous release of A1 pulley release will be performed in the well-managed operation theater set up, using an 18 gauge hypodermic needle, after preparation of the skin and injection of 1ml 2% plain lidocaine. The proper location of the pulley will be defined using surface landmarks in each digit after waiting a few minutes to allow the anesthetic to take effect the 18 gauge needle will be longitudinally moved to keep the level of the needle parallel with the tendon grating sensation will be elucidated confirming the cut of pulley until there is no grating sensation felt and improvement of symptoms. A sterile dressing will be placed.
  Arms: percutaneous release

SUMMARY:
Trigger fingers (TF) is the common cause of pain and disturbed function of hand. Many studies show that percutaneous release of A1 pulley has better outcome than the steroid injection. However, over the past many years, steroid injection has been considered as the choice of treatment after the failure of conservative treatment methods. The aim of this study is to assess the effect of percutaneous release of A1 pulley compared with the local Steroid injection in the treatment of trigger fingers.

This study is based on a randomized clinical trial to compare the effect of the percutaneous release of A1 pulley with steroid injection in trigger fingers. A total of 112 participants aged 18 years and above suffering from trigger fingers with failed conservative treatment will be intervened randomly (56 participants in injection group and 56 participants in percutaneous release group). The Quinnell's classification, VAS scoring system and active range of movement in the affected site will be assessed at the baseline and the same criteria will be at one month and three month as end line assessment. Statistical analyses will be performed using independent t-test and Mann Whitney U test to compare between the two means. The outcome of this study will help to guide the physicians to choose the better therapeutic approach among the patients suffering from trigger fingers.

DETAILED DESCRIPTION:
Stenosing flexor tenosynovitis also known as trigger finger. It is a common clinical condition where there is locking and clicking during flexion and extension of the involved digit or even locking. The trigger ring finger is the first commonest, and the trigger thumb is the second commonest of trigger fingers. Flexor tendon gliding motion is dependent on a 'Critical Tendon Sheath Caliber Tolerance' which allows passage of flexor tendon through the A1 pulley in the Metacarpophalangeal joint.

The prevalence of trigger finger is 2 % in the general population, which is most common in women in the fifth or sixth decade of life. The possibility of a trigger finger is between 2 and 3% during the lifetime, which increases up to 10 % in diabetic patients. The trigger finger in diabetic patients suffered from worse renal function and glycemic control, along with a higher incidence of cardiovascular disease. The causes of Trigger finger are still not well known, some factors may increase the risk of developing the condition such as forceful hand activities (mechanical irritation, congenital and medical conditions (Diabetes and Rheumatoid arthritis). Trigger thumb is caused by thickening of flexor tendon gliding at the tendon A1 pulley interface or thickening of A1 pulley.

Diagnosis is primarily made based on physical examination. The patients often present with pain or clicking at the metacarpal head, which causes difficulty in holding or grasping objects. In most advanced cases, there is locking in flexion or extension position.

Nowadays, the morphological changes in the case of trigger fingers can be ruled out by high-resolution ultrasonography with a high-frequency transducer, and it has been found that the cut-off for pathological findings is a 20% increase in tendon thickness compared to the contralateral tendon. The average width and thickness of the A1 pulley are 7.1 mm and less than 1 mm respectively.

Treatment of Trigger fingers includes conservative such as splinting, oral medications, injection, and surgical management such as open release, and percutaneous release. Steroid injection has been serving us as a traditional way of injection therapy for many years for those who are not getting better with oral medications and physiotherapy. Steroid injection is effective because of its anti-inflammatory properties.

The first percutaneous release was performed in 1958 and the success rate was 100% without any reported complications. Percutaneous A1 pulley release has been the method of choice for patients who does not respond to conservative treatment (local steroid) with low complication rates.

There is a concern regarding percutaneous release in the thumb, where tendon sheath and neurovascular bundle are in proximity.

The technique of local steroid injection into the flexor sheath was described by Howard in 1953. It has become an accepted initial treatment for trigger fingers largely due to its use within the outpatient department and its low complication rate.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged 18 years and above
* Duration of symptoms :≥ 3 months
* Triggering in any of the digits of hand
* Trigger finger type II-IV based on Quinnell classification

Exclusion Criteria:

* There is prior treatment for trigger finger, or Trigger thumb
* There had been previous surgery or other hand pathology such as rheumatoid arthritis, osteoarthritis, Dupuytren's contracture and diabetic mellitus.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-11-02 (Actual); Study Completion 2022-11-02 (Actual)

PRIMARY OUTCOMES:
Functional mobility improvement | 3 months
  Compare the effects of percutaneous release versus steroid injection on functional mobility at baseline, one month and three months.
Pain reduction | 3 months
  Compare the effects of percutaneous release versus steroid injection on pain reduction at baseline, one month and three months.

SECONDARY OUTCOMES:
Decrease in the thickness of the A1 pulley | 3 months
  Compare the effects of percutaneous release versus steroid injection on decrease in the thickness at baseline, one month and three months.
Recurrence of problem within 3 months | 3 months
  Compare the effects of percutaneous release with steroid injection on problem recurrence in three months.

CONTACTS AND LOCATIONS:
Overall Officials: Mandeep Karki, MS, Principal Investigator — Nepal Orthopedic Hospital
Locations (1):
- Armed Police Force Hospital, Kathmandu, Bagmati, Nepal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Moore JS. Flexor tendon entrapment of the digits (trigger finger and trigger thumb). J Occup Environ Med. 2000 May;42(5):526-45. doi: 10.1097/00043764-200005000-00012. PMID 10824306
- [Result] Maneerit J, Sriworakun C, Budhraja N, Nagavajara P. Trigger thumb: results of a prospective randomised study of percutaneous release with steroid injection versus steroid injection alone. J Hand Surg Br. 2003 Dec;28(6):586-9. doi: 10.1016/s0266-7681(03)00172-4. PMID 14599834
- [Result] Makkouk AH, Oetgen ME, Swigart CR, Dodds SD. Trigger finger: etiology, evaluation, and treatment. Curr Rev Musculoskelet Med. 2008 Jun;1(2):92-6. doi: 10.1007/s12178-007-9012-1. PMID 19468879
- [Result] Mineoka Y, Ishii M, Hashimoto Y, Yuge H, Toyoda M, Nakamura N, Katsumi Y, Fukui M. Trigger finger is associated with risk of incident cardiovascular disease in individuals with type 2 diabetes: a retrospective cohort study. BMJ Open Diabetes Res Care. 2021 Apr;9(1):e002070. doi: 10.1136/bmjdrc-2020-002070. PMID 33832915
- [Result] David M, Rangaraju M, Raine A. Acquired triggering of the fingers and thumb in adults. BMJ. 2017 Nov 30;359:j5285. doi: 10.1136/bmj.j5285. No abstract available. PMID 29191846
- [Result] Lunsford D, Valdes K, Hengy S. Conservative management of trigger finger: A systematic review. J Hand Ther. 2019 Apr-Jun;32(2):212-221. doi: 10.1016/j.jht.2017.10.016. Epub 2017 Dec 28. PMID 29290504
- [Result] Takahashi M, Sato R, Kondo K, Sairyo K. Morphological alterations of the tendon and pulley on ultrasound after intrasynovial injection of betamethasone for trigger digit. Ultrasonography. 2018 Apr;37(2):134-139. doi: 10.14366/usg.17038. Epub 2017 Jul 25. PMID 28870061
- [Result] Pan M, Sheng S, Fan Z, Lu H, Yang H, Yan F, E Z. Ultrasound-Guided Percutaneous Release of A1 Pulley by Using a Needle Knife: A Prospective Study of 41 Cases. Front Pharmacol. 2019 Mar 26;10:267. doi: 10.3389/fphar.2019.00267. eCollection 2019. PMID 30971922
- [Result] Bianchi S, Gitto S, Draghi F. Ultrasound Features of Trigger Finger: Review of the Literature. J Ultrasound Med. 2019 Dec;38(12):3141-3154. doi: 10.1002/jum.15025. Epub 2019 May 20. PMID 31106876
- [Result] LORTHIOIR J Jr. Surgical treatment of trigger-finger by a subcutaneous method. J Bone Joint Surg Am. 1958 Jul;40-A(4):793-5. No abstract available. PMID 13549516
- [Result] Blumberg N, Arbel R, Dekel S. Percutaneous release of trigger digits. J Hand Surg Br. 2001 Jun;26(3):256-7. doi: 10.1054/jhsb.2001.0569. PMID 11386779
- [Result] Park MJ, Oh I, Ha KI. A1 pulley release of locked trigger digit by percutaneous technique. J Hand Surg Br. 2004 Oct;29(5):502-5. doi: 10.1016/j.jhsb.2004.03.015. PMID 15336757
- [Result] Ragoowansi R, Acornley A, Khoo CT. Percutaneous trigger finger release: the 'lift-cut' technique. Br J Plast Surg. 2005 Sep;58(6):817-21. doi: 10.1016/j.bjps.2005.04.003. PMID 15936736
- [Result] Eastwood DM, Gupta KJ, Johnson DP. Percutaneous release of the trigger finger: an office procedure. J Hand Surg Am. 1992 Jan;17(1):114-7. doi: 10.1016/0363-5023(92)90125-9. PMID 1538091
- [Result] Lyu SR. Closed division of the flexor tendon sheath for trigger finger. J Bone Joint Surg Br. 1992 May;74(3):418-20. doi: 10.1302/0301-620X.74B3.1587893.
- [Result] Bain GI, Turnbull J, Charles MN, Roth JH, Richards RS. Percutaneous A1 pulley release: a cadaveric study. J Hand Surg Am. 1995 Sep;20(5):781-4; discussion 785-6. doi: 10.1016/S0363-5023(05)80430-7. PMID 8522744
- [Result] HOWARD LD Jr, PRATT DR, BUNNELL S. The use of compound F (hydrocortone) in operative and non-operative conditions of the hand. J Bone Joint Surg Am. 1953 Oct;35-A(4):994-1002. No abstract available. PMID 13108902
- [Result] Dala-Ali BM, Nakhdjevani A, Lloyd MA, Schreuder FB. The efficacy of steroid injection in the treatment of trigger finger. Clin Orthop Surg. 2012 Dec;4(4):263-8. doi: 10.4055/cios.2012.4.4.263. Epub 2012 Nov 16. PMID 23205235
- [Result] Wang J, Zhao JG, Liang CC. Percutaneous release, open surgery, or corticosteroid injection, which is the best treatment method for trigger digits? Clin Orthop Relat Res. 2013 Jun;471(6):1879-86. doi: 10.1007/s11999-012-2716-6. Epub 2012 Dec 4. PMID 23208122
- [Result] Quinnell RC. Conservative management of trigger finger. Practitioner. 1980 Feb;224(1340):187-90. No abstract available. PMID 7367373
- [Result] Sato ES, Gomes Dos Santos JB, Belloti JC, Albertoni WM, Faloppa F. Treatment of trigger finger: randomized clinical trial comparing the methods of corticosteroid injection, percutaneous release and open surgery. Rheumatology (Oxford). 2012 Jan;51(1):93-9. doi: 10.1093/rheumatology/ker315. Epub 2011 Oct 29. PMID 22039269
- [Result] Sahu R, Gupta P. Experience of Percutaneous Trigger Finger Release under Local Anesthesia in the Medical College of Mullana, Ambala, Haryana. Ann Med Health Sci Res. 2014 Sep;4(5):806-9. doi: 10.4103/2141-9248.141558. PMID 25328798
- [Result] Ha KI, Park MJ, Ha CW. Percutaneous release of trigger digits. J Bone Joint Surg Br. 2001 Jan;83(1):75-7. doi: 10.1302/0301-620x.83b1.11247. PMID 11245542
- [Result] Saldana MJ. Trigger digits: diagnosis and treatment. J Am Acad Orthop Surg. 2001 Jul-Aug;9(4):246-52. doi: 10.5435/00124635-200107000-00004. PMID 11476534
- [Derived] Karki M, Sharma R, Sunuwar DR, Gupta RS, Singh DR, Lama S, Bhandari KK, Tamang RK, Chaudhary NK. Effect of percutaneous release versus steroid injection among adults with trigger fingers: a randomized clinical trial. BMC Musculoskelet Disord. 2025 Oct 1;26(1):885. doi: 10.1186/s12891-025-08981-6. PMID 41029287